CLINICAL TRIAL: NCT02374970
Title: Effectiveness of Transversus Abdominis Muscular Training in Patients With Chronic Low Back Pain
Brief Title: Transversus Abdominis Muscular Training and Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P14/084
Record Dates: First submitted 2015-02-19; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Actual Lumbar stability exercises involving co-contraction of the transversus abdominis and Protocolized Physiotherapy (therapeutic exercises and thermotherapy during 12 sessions)
  Interventions: Other: Lumbar stability exercises; Other: Protocolized Physiotherapy
- Control group (Active Comparator): Protocolized Physiotherapy treatment: therapeutic exercises and thermotherapy during 12 sessions.
  Interventions: Other: Protocolized Physiotherapy

INTERVENTIONS:
Other: Lumbar stability exercises — Four individualized learning sessions will be held during the same period of protocolized physiotherapy. Biofeedback training using the ultrasound machine will be performed in the first session, in order to show the specific contraction of the abdominal muscles with the stability exercises. The other three learning sessions will be performed without feedback, for the patient learn the exercises to make at home during the follow-up period.
  Arms: Intervention group
Other: Protocolized Physiotherapy — Therapeutic exercises and thermotherapy during 12 daily sessions

SUMMARY:
Low back pain is not a diagnosis; it is a symptom describing the presence of pain in the lumbar vertebral or paravertebral region without any reference to the structure or cause of the process. It is one of the most widespread diseases and one of the most common reasons for visits in primary care setting.

Exercises to improve lumbar stability involving co-contraction of the transversus abdominis have proved to be effective in reducing pain and improving function. It has been stated by ultrasound images that specific stabilization exercises cause contraction of the deep abdominal muscles, but it remains unclear whether training produce thickness muscle improvement and if this improvement is related to clinical findings.

To try to resolve this issue a project of an experimental trial, double-blind (patient and evaluator) with two groups randomly assigned is presented. All participants will be recruited in an primary care center of the Catalan Health Institut and will sign informed consent. All will receive a protocolized treatment with therapeutic exercises and thermotherapy and, additionally, those assigned to the intervention group were instructed in performing lumbar stability exercises.

Pain (VAS), function (Roland-Morris Questionnaire) and the thickness of the transversus abdominis, internal and external oblique muscles (measured by ultrasound) at baseline, end of treatment protocol (12 sessions) and three months after the end of treatment will be assessed.

Results in pain, function, and its correlation with the mean changes in the thickness of transversus abdominis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Diagnosis of chronic low back pain (over 3 months)
* Sign the informed consent form.

Exclusion Criteria:

* Non-stand supine position
* Neural Irradiation pain
* Previous surgical intervention in low back region
* Heart pathology
* Pregnancy
* Pending litigation or legal claim
* Poor language and communication skills making difficult to understand the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in transversus abdominis muscle thickness (Ultrasonography) | Baseline, 15 days after, and three months after

SECONDARY OUTCOMES:
Change in pain intensity (Visual analogue scale) | Baseline, 15 days after, and three months after
Disability (Roland-Morris questionnaire) | Baseline, 15 days after, and three months after
Change in internal oblique muscle thickness (Ultrasonography) | Baseline, 15 days after, and three months after
Change in external oblique muscle thickness (Ultrasonography) | Baseline, 15 days after, and three months after
Patient perception of change (Global Rating of Change scale) | 15 days after recruitment, and three months after

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Villar-Mateo, Principal Investigator — Jordi Gol Institut of Research in Primary Health Care
Locations (1):
- Catalan Health Institut. Sant Ildefons Rehabilitation Service, Cornellà de Llobregat, Barcelona, Spain